CLINICAL TRIAL: NCT02412033
Title: Vaginal Misoprostol Prior to Intrauterine Contraceptive Device Insertion in Women With Previous Caesarean Section
Brief Title: Misoprostol Prior to Intrauterine Contraceptive Device Insertion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamad sayed abdellah, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IUD- CS
Record Dates: First submitted 2015-04-04; First posted 2015-04-08 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pain Prior to IUD Insertion
Keywords: vaginal misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol group (Active Comparator): Going to receive 400 µg misoprostol vaginally 3 hours before IUD insertion.
  Interventions: Drug: Misoprostol
- Placebo group (Placebo Comparator): Going to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 400 µg misoprostol vaginally 3 hours before IUD insertion.
  Arms: Misoprostol group
Drug: Placebo — This group will receive placebo
  Arms: Placebo group

SUMMARY:
Intrauterine devices (IUDs) are widely used as reversible contraceptives. Both copper- and levonorgestrel (LNG)-releasing IUDs (LNG-IUDs) are safe,cost-effective in the long term and equally effective compared with tubal sterilization.

In addition, the LNG-IUD (Mirena®) provides non contraceptive benefits, such as treatment for menorrhagia, dysmenorrhea and anemia. The current use of IUDs among reproductive-aged women ranges from 8 to 15% worldwide. Reported complications related to IUD insertion are 8.8% insertion failure, 2.8-11.5% cervical problems, 0.2% cervical perforation, 0.2% syncope and 5.8% expulsion. Insertion failures and cervical problems seem to occur more often among women who have never delivered vaginally.

Cervical stenosis, an immature or small cervix and a significantly ante- or retroverted position of the uterus, has been described as factors associated with a difficult sounding of the cervical canal or even failure to insert the IUD.

Misoprostol is an inexpensive prostaglandin E1-analogue, which is associated with few side effect. More over several have shown the benefit of misoprostol as a cervical ripening agent in non pregnant women. Priming with misoprostol prior to hysteroscopy and dilatation and curettage (D&C) in perimenopausal women resulted in increased cervical dilatation and lower rate of cervical laceration.

The effect of misoprostol on the cellular matrix causes dissolution of collagen fiber increasing the amount of fluid in the stroma and consequentially causes cervical effacement. Fear of pain during insertion, however, might prevent some women from choosing IUD and fears of painful and/or difficult placements may lead them to recommend or counsel women on other, less effective methods.

Women's perception of pain is multifactorial and likely to be influenced by cultural differences and personal experiences; insertion-related pain is therefore difficult to predict. Nevertheless, factors associated with greater pain include nulliparity, not currently breastfeeding and longer time since last pregnancy; of these factors, nulliparity is the strongest predictor of pain.

The proportion of women of reproductive age who are nulliparous is increasing, with women delaying childbirth and having fewer children or choosing to remain childless. The proportion of Caesarean section births has also increased and women who have only ever had a Caesarean section are often viewed as nulliparous with respect to IUD placement. Anticipated pain is often greater than the actual pain experienced, and the majority of nulliparous women experience no more than moderate pain during IUD insertion. However, among nulliparous women there is a subset (about 17%) for whom the insertion of IUD is associated with severe pain.These women need effective pain relief.

For most nulliparous, nulligravid or parous women, IUD insertion can be performed successfully without cervical priming and with a minimum amount of discomfort. Whether selective use of misoprostol has a role in management of pain in certain subsets of women (e.g. nulliparous women and those in whom the insertion is non-routine/difficult) has yet to be adequately studied.

ELIGIBILITY:
Inclusion Criteria:

1. Include those who delivered by CS .
2. Who accept to participate in the study.
3. Desire IUD placement.
4. Negative pregnancy test.
5. No history or current history of pelvic inflammatory disease.
6. No current cervicitis.
7. No contraindication to IUD insertion (less than 4 week post partum,gynecological malignancy,unexplained vaginal bleeding and pregnancy).

Exclusion Criteria:

1. Any contraindication to IUD .
2. Current pregnancy.
3. Uterine anomaly.
4. Undiagnosed abnormal uterine bleeding.
5. Allergy to misoprostol.
6. Patients contraindicated to administration of misoprostol.
7. Women who delivered vaginally.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
easiness score of IUD insertion | 5 minutes

SECONDARY OUTCOMES:
the difference in the pain intensity scores between the study groups | 5 minutes
the women's level of satisfaction at the end of insertion | 5 minutes

IPD SHARING:
Plan to Share IPD: Undecided